CLINICAL TRIAL: NCT02077270
Title: Pretreatment With Electroacupuncture to Reduce Discomfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dan Carter, Gastroenterologist, GI consult, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SHEBA-14-9733-DC-CTIL
Record Dates: First submitted 2014-02-24; First posted 2014-03-04 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pain
Keywords: colonoscopy; acupuncture; pain
MeSH Terms: conditions — Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- electroacupuncture (Experimental): patients in whom precolonoscopic electroacupuncture is preformed
  Interventions: Procedure: electroacupuncture
- Sham electroacupuncture (Placebo Comparator): sham electroacupuncture
  Interventions: Procedure: electroacupuncture
- No intervantion (Sham Comparator): no intervantion
  Interventions: Procedure: electroacupuncture

INTERVENTIONS:
Procedure: electroacupuncture — Patients allocated to this arm will receive electro-acupuncture bilaterally on the following points which are considered relevant both for sedation and abdominal distention:LI4 (Hegu),ii. St36 (Zusanli), Sp6 (Sanyinjiao), St25 (Tianshuv),. Du20 (Baihui),

SUMMARY:
The main hypothesis is that performance of electroacupuncture before colonoscopy reduces pain during the exam.

DETAILED DESCRIPTION:
To assess the efficacy of pre-colonoscopic electroacupuncture in reducing discomfort during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients referred for their first colonoscopy in the department of GI in Sheba, Tel Hashomer

Exclusion Criteria:

1. Ages <18y >75y
2. Any prior gastrointestinal endoscopy.
3. History of colonic resection.
4. Known or suspected stenosis of the colon.
5. Pregnancy.
6. Inflammatory bowel disease
7. Neuropsychiatric disorders or receiving psychotropic drugs.
8. Prior knowledge or experience of acupuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of pre-colonoscopic electroacupuncture in reducing discomfort during colonoscopy by measuring sedative drug amounts during colonoscopy | during the colonoscopy and in the hour post procedure
  The measurement of the amount of drug added during colonoscopy

SECONDARY OUTCOMES:
Time of insertion till the cecum. | during colonoscopy
  Time between insertion of the colonoscopy and the image of the cecum
Time of post-colonoscopy recovery as measured by the Aldrete score | up to 1 hour post colonoscopy
Number of intra-examination adverse events. | from the begining of the endoscopy and up to 1 hour post procedure
Patient's total satisfaction with the exam and the analgesia | between the end of the procedure and up to 1 hour post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel